CLINICAL TRIAL: NCT04020627
Title: Acute Effects of BIPAP vs CPAP on Hemodynamics and Respiratory Parameters in Management of Type 2 Respiratory Failure Patients
Brief Title: BIPAP vs CPAP Effects on Type 2 Respiratory Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Shabana Kausar
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Respiratory Failure
Keywords: Respiratory failure; BiPap; CPap; Respiratory Parameters; Hemodynamics
MeSH Terms: conditions — Hypoventilation; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BiPAP Group (Experimental): Bilevel Positive Airway Pressure
  Interventions: Other: BiPAP Group
- CPAP Group (Experimental): Continuous Positive Airway Pressure
  Interventions: Other: CPAP Group

INTERVENTIONS:
Other: BiPAP Group — BIPAP
  - 1hr after every 6hrs for 3 days/week Conventional physiotherapy Treatment (Percussion, vibration, shaking) Modified postural drainage Incentive spirometer Blow bottle/Tissue blowing/Positive Expiratory Pressure(PEP) device
  Arms: BiPAP Group
Other: CPAP Group — CPAP
  - 1hr after every 6hrs for 3 days/week Conventional physiotherapy Treatment (Percussion, vibration, shaking) Modified postural drainage Incentive spirometer Blow bottle/Tissue blowing/PEP device
  Arms: CPAP Group

SUMMARY:
Effectiveness of BIPAP is evaluated in Type-2 failure but evaluation of effectiveness of CPAP in Type-2 respiratory failure in post cardiac surgery patients was not done. So the objective of this study is to determine the acute effects of BIPAP vs. CPAP with conventional physiotherapy on Hemodynamics and Respiratory parameters in management of Type 2 Respiratory failure in post cardiac surgery patients.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) refers to the provision of Ventilatory support through the patient's upper airway using a mask or similar device. This technique is distinguished from those which bypass the upper airway with a tracheal tube, laryngeal mask, or tracheotomy and are therefore considered invasive. NIV refers to non-invasive positive pressure ventilation, Continuous positive airway pressure (CPAP) refers to the non-invasive application of positive airway pressure, again using a face or nasal mask rather than in conjunction with invasive techniques.

A study on Non-invasive ventilation in postoperative patients was conducted in 2017 in Italy; systematic review was performed on Patients undergoing any of the following procedures, thoracic surgery, lung surgery, abdominal surgery, solid organ transplantation, thoraco-abdominal surgery and bariatric surgery were included. Information on demographics, medical history, preoperative medications, postoperative care Pharmacologic management and laboratory investigation results were obtained from medical charts.

Prospective, randomized, case-controlled, pilot study included forty patients, who underwent elective (OPCAB) and were randomized into two groups. group-A (BiPAP) and group-B . All patients received same regimen of medication. Group-B was kept on BiPAP immediately following extubation, while, group-B received conventional physiotherapy only. All hemodynamic and oxygenation parameter were recorded and chest radiographs were done to find out incidence of atelectasis. Patients were followed up to their discharge.

Noninvasive Ventilatory support does not facilitate recovery from acute respiratory failure in chronic obstructive pulmonary disease his investigation evaluates, in a prospective, randomized and controlled manner, whether noninvasive ventilatory support (NIVS) with bilevel positive airway pressure (BiPAP) facilitates recovery from acute respiratory failure (ARF) in patients with chronic obstructive pulmonary disease.

Effects of Positive Airway Pressure in Patients with Heart Failure and Obstructive Sleep Apnea done at Toronto General Hospital University Health Network and Mount Sinai Hospital Twenty-four patients with a depressed left ventricular ejection fraction (45 percent or less) and obstructive sleep apnea who were receiving optimal medical treatment for heart failure underwent polysomnography. The subjects were then randomly assigned to receive medical therapy either alone (12 patients) or with the addition of continuous positive airway pressure (12 patients) for one month. The assessment protocol was then repeated.

Bilevel positive airway pressure on ventricular ectopy in heart failure patients with obstructive sleep apnoea was done at canada in 2015. Following optimisation of medical treatment and cpap.The frequency of vpbs and urinary norepinephrine (noradrenaline) concentrations during total sleep time were determined at baseline and after 1 month

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 respiratory Failure partial pressure of Oxygen(PaO2) of <8 kilopascal(kPa) and pco2 of >6 kpa with a respiratory acidosis pH<7.35 (H+>45nmol/L) guidelines provided by British Thoracic society.
* Patients with Sleep apnea /acute confusional state (Psychosis)

Exclusion Criteria:

* Person with Surgical Emphysema
* Pneumothorax
* Medically unstable (hypotensive shock, uncontrolled cardiac ischemia, or arrhythmia
* Person with Bulla's disease
* Severe bronchospasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Arterial blood gas (ABG) parameter like potential of hydrogen (PH) | 3rd Day
  Above parameter was measured by serial ABG analysis. Its normal reference range is 7.35-7.45. baseline reading will be taken at 10 minutes before starting Non invasive ventilation training. Changes from the Baseline
Arterial blood gas parameter like bicarbonate(HCO3). | 3rd Day
  Above parameter was measured by serial ABG analysis. Its normal reference range is 22-28 nmol/L. Baseline reading will be taken at 10 minutes before starting Non invasive ventilation training. Changes from the Baseline
Arterial blood gas parameter like partial pressure of carbon dioxide (PCO2) | 3rd Day
  Above parameter was measured by serial ABG analysis. Its normal reference range is 35-45 mmHg. Baseline reading will be taken at 10 minutes before starting Non invasive ventilation training. Changes from the Baseline
Arterial blood gas parameter like partial pressure of carbon dioxide (PO2) | 3rd Day
  Above parameter was measured by serial ABG analysis. Its normal reference range is 80-100 mmHg. Baseline reading will be taken at 10 minutes before starting Non invasive ventilation training. Changes from the Baseline
Heart Rate | 3rd Day
  Changes from the Baseline, It will be measured through Cardiac Monitor
Saturation (SPO2) | 3rd Day
  Changes from the Baseline, It will be measured in percentage through Cardiac Monitor.
Systolic Blood Pressure (SBP) | 3rd day
  Changes from the Baseline, It was measure through sphygmomanometer and Blood pressure is measured in units of millimeters of mercury (mmHg). The readings are always given in pairs, with the upper (systolic) value first, followed by the lower (diastolic) value.
Diastolic Blood Pressure (SBP) | 3rd Day
  Changes from the Baseline, It was measure through sphygmomanometer and Blood pressure is measured in units of millimeters of mercury (mmHg). The readings are always given in pairs, with the upper (systolic) value first, followed by the lower (diastolic) value.

SECONDARY OUTCOMES:
Richmond Agitation-Sedation Scale (RASS) | 3rd day
  Richmond Agitation-Sedation Scale is a medical scale used to assess the agitation or sedation level of a individual. Changes from the Baseline. Below 0 means drowsy and sedated, 0 means alert and calm and 1 or above 1 means restless & agitated
Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) | 3rd Day
  Changes from the baseline. It will provide a qualitative result of "delirium present" or "delirium absent". Clinical psychologist delirium is defined in terms of four diagnostic features, and is deemed present when a patient has positive Feature 1 and Feature 2 and either Feature 3 or 4. overall answer in Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] British Thoracic Society Standards of Care Committee. Non-invasive ventilation in acute respiratory failure. Thorax. 2002 Mar;57(3):192-211. doi: 10.1136/thorax.57.3.192. No abstract available. PMID 11867822
- [Background] Antonelli M, Conti G, Rocco M, Bufi M, De Blasi RA, Vivino G, Gasparetto A, Meduri GU. A comparison of noninvasive positive-pressure ventilation and conventional mechanical ventilation in patients with acute respiratory failure. N Engl J Med. 1998 Aug 13;339(7):429-35. doi: 10.1056/NEJM199808133390703. PMID 9700176
- [Background] Pelosi P, Severgnini P, Aspesi M, Gamberoni C, Chiumello D, Fachinetti C, Introzzi L, Antonelli M, Chiaranda M. Non-invasive ventilation delivered by conventional interfaces and helmet in the emergency department. Eur J Emerg Med. 2003 Jun;10(2):79-86. doi: 10.1097/00063110-200306000-00002. PMID 12789060
- [Background] Pieczkoski SM, Margarites AGF, Sbruzzi G. Noninvasive Ventilation During Immediate Postoperative Period in Cardiac Surgery Patients: Systematic Review and Meta-Analysis. Braz J Cardiovasc Surg. 2017 Jul-Aug;32(4):301-311. doi: 10.21470/1678-9741-2017-0032. PMID 28977203
- [Background] Mehta Y, Vats M, Kumar SK, Singh S, Khurana P, Trehan N. Prevention of postoperative atelectasis in the post-cardiac surgical patient with poor left ventricular function: A study of the efficacy of Bi-level positive airway pressure. Chest. 2017 Oct 1;132(4):537A
- [Background] Olper L, Bignami E, Di Prima AL, Albini S, Nascimbene S, Cabrini L, Landoni G, Alfieri O. Continuous Positive Airway Pressure Versus Oxygen Therapy in the Cardiac Surgical Ward: A Randomized Trial. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):115-121. doi: 10.1053/j.jvca.2016.08.007. Epub 2016 Aug 10. PMID 27771274
- [Background] Barbe F, Togores B, Rubi M, Pons S, Maimo A, Agusti AG. Noninvasive ventilatory support does not facilitate recovery from acute respiratory failure in chronic obstructive pulmonary disease. Eur Respir J. 1996 Jun;9(6):1240-5. doi: 10.1183/09031936.96.09061240. PMID 8804944
- [Background] Kaneko Y, Floras JS, Usui K, Plante J, Tkacova R, Kubo T, Ando S, Bradley TD. Cardiovascular effects of continuous positive airway pressure in patients with heart failure and obstructive sleep apnea. N Engl J Med. 2003 Mar 27;348(13):1233-41. doi: 10.1056/NEJMoa022479. PMID 12660387